CLINICAL TRIAL: NCT04403932
Title: Cohort Study to Determine the Association Between Vitamin D Deficiency and Severity of the Disease in Patients With Coronarvirus Disease 2019 (COVID-19)
Brief Title: Increased Risk of Severe Coronavirus Disease 2019 in Patients With Vitamin D Deficiency
Acronym: COVIT-D
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Fernando Macaya, MD, Hospital San Carlos, Madrid
Other Study IDs: 20/428-E_COVID
Record Dates: First submitted 2020-05-24; First posted 2020-05-27 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: Coronavirus Disease 2019 (COVID-19); Vitamin D Deficiency; Severe Acute Respiratory Syndrome; Angiotensin Converting Enzyme 2
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective observational study we aim to study the association of vitamin D deficiency with adverse clinical outcomes in patients infected with Coronavirus disease 2019

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) can induce an exaggerated inflammatory response. Vitamin D is a key modulator of the immune system. We hypothesized that vitamin D deficiency (VDD) could increase the risk of developing severe COVID-19 infection. The COVIT-D study (Increased risk of severe COVID-19 infection in patients with Vitamin D deficiency) is a prospective cohort study recruiting patients with confirmed COVID-19 seen at the emergency department of a tertiary hospital. A measurement of 25-hydroxyvitamin D is obtained at admission and follow-up obtained. The primary outcome is a composite of death, admission to the intensive care unit, and/or a need for higher oxygen flow than that provided by nasal cannula. The primary association between VDD - categorised in groups - and the primary outcome will be evaluated with univariate analyses and multivariable logistic regression including the following prespecified confounders: age, gender, obesity and chronic kidney disease. The estimated sample size is n=500 and the expected inclusion time lapse 3 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* symptoms suggestive of COVID-19
* positive reverse-transcriptase polymerase chain reaction or antibodies for SARS-CoV-2

Exclusion Criteria:

* Bacterial community acquired pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult subjects attending the emergency department with symptoms suggestive of COVID-19 and a positive reverse-transcriptase polymerase chain reaction for SARS-CoV-2
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
severe COVID-19 | 17/04/2020 to 01/06/2020
  death, admission to the intensive care unit, and/or a need for higher oxygen flow than that provided by nasal cannula

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain